CLINICAL TRIAL: NCT04074720
Title: Prospective Breast Cancer Biospecimen Collection
Status: Recruiting | Type: Observational
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Other Study IDs: 16D.674; JT 8877 (Other: JeffTrial Number)
Record Dates: First submitted 2019-08-01; First posted 2019-08-30 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer; Invasive Breast Cancer; Carcinoma in Situ of the Breast
Keywords: Breast Cancer; Tumor Tissue Collection; Serum Collection; Plasma Collection; Fresh Tissue Collection; Fixed Tissue Collection; Translational Research; Biospecimen Collection; Surgical Resection; Vascular Access Placement
MeSH Terms: conditions — Breast Neoplasms; Breast Carcinoma In Situ

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumor and normal adjacent tissue samples will be collected from approximately 200 living patients with breast cancer irrespective of hormone status under the care of TJUH clinicians. Serum will be collected at the same time as serum and adjacent normal so that serum exosomes as well as extracellular matrix influences can be examined.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group 1: Newly Diagnosed Breast Cancer Patients: Tissue will be procured during a standard of care procedure the patient will already have scheduled. A one time blood draw will be performed at this time and an optional rectal swab for biome analysis may occur. Follow up will only consist of chart review to determine date of recurrence, metastases, and/or death.
  Interventions: Procedure: Tissue Sample collection; Other: Blood Sample Collection; Other: Rectal Swab
- Group 2: Patients with Brain Metastases from Primary Breast Cancer: The brain metastasis specimen experiments will use tissue from 36 patients (12 per subtype: estrogen positive, Her-neu-2 positive, and triple negative). Tissue will be procured during a standard of care procedure the patient will already have scheduled. A one time blood draw will be performed at this time and an optional rectal swab for biome analysis may occur. Follow up will only consist of chart review to determine date of recurrence, metastases, and/or death.
  Interventions: Procedure: Tissue Sample collection; Other: Blood Sample Collection; Other: Rectal Swab

INTERVENTIONS:
Procedure: Tissue Sample collection — Tissue sample collected following standard of care procedure patient was already scheduled to have
Other: Blood Sample Collection — A one time sample of blood will be collected on day of standard of care procedure
Other: Rectal Swab — optional rectal swab may be collected on day of standard of care procedure

SUMMARY:
Tissue will be procured during a standard of care procedure the patient will already be scheduled to undergo. A one time blood draw will be performed at this time and an optional rectal swab for biome analysis may occur. Follow Up will only consist of chart review to determine date of recurrence, metastases, and/or death

DETAILED DESCRIPTION:
This is a breast cancer biospecimen and possible metastasis procurement study with the goal of obtaining specimens appropriately for genomic and proteomic analysis. Other than reviewing and signing the consent form by the participants in the study, and the study-specific blood tissue procurement and blood draw (and optional biome specimen), all care and clinical encounters will be as per standard of care. There are four times when tissue may be procured and an optional biome specimen collection depending on the treatment course the treating team decides upon. The technique will be chosen based on physician discretion, patient medical treatment, and patient preference. Treatment regimen will consist of tumor sampling/extraction, one blood draw, optional biome specimen collection, and sample storing. This is a single arm study; all participants will have tissue and blood sample procured for biospecimen analysis and repository. Patients have the option to donate a biome specimen as well. Providing the biome sample is optional and will not influence eligibility to patient participation in this study. There will be no assignment or randomization to different treatment groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years old at time of consent
* Subject must be capable to giving informed consent or have an acceptable surrogate capable of giving consent on the subject behalf.
* Patients with carcinoma in situ or invasive breast cancer
* Patient must be undergoing one of the following:

  * definitive surgical tumor resection for breast cancer OR
  * placement of a vascular access device as a prelude to neoadjuvant therapy for breast cancer OR
  * neurosurgical resection of a brain metastasis from primary breast cancer.

Exclusion Criteria:

* <18 years old
* Not able to give informed consent and does not have acceptable surrogate capable to giving informed consent.
* Active drug/alcohol dependence or abuse history

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults (≥18 years old) with newly diagnosed in situ carcinoma or invasive breast cancer, or patients with primary breast cancer with metastasis to the brain. Up to 200 newly diagnosed breast cancer patients, and 36 patients with brain metastases.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2018-05-10 (Actual); Primary Completion 2028-07-01 (Estimated); Study Completion 2028-07-01 (Estimated)

PRIMARY OUTCOMES:
Tumor biomarker identification | Up to 5 years
  Collected biospecimens will be analyzed using current laboratory techniques to identify the presence of breast cancer biomarkers such as estrogen receptor (ER) and human epidermal growth factor receptor 2 (HER2).

SECONDARY OUTCOMES:
Laboratory-based breast cancer tumor genomic profile | Up to 5 years
  Genomic profile will be based on laboratory analysis of the collected tumor tissue biospecimens to identify how genes interact with the tumor and its environment.

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Simone, MD, Principal Investigator — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (1):
- Sidney Kimmel Cancer Center at Thomas Jefferson University, Philadelphia, Pennsylvania, United States